CLINICAL TRIAL: NCT04460859
Title: RecruitmEnt Assessed by eleCtRical Impedance Tomography: Feasibility, Correlation With Clinical oUtcomes and pIloT Data on Personalised PEEP Selection.
Brief Title: RecruitmEnt Assessed by eleCtRical Impedance Tomography
Acronym: RECRUIT
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 2027
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Mechanical Ventilation; Lung recruitment; ARDS; Electrical impedance tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intubated mechanically ventilated ARDS patients: Intubated mechanically ventilated patients with moderate to severe ARDS according to the Berlin definition
  Interventions: Other: Specific lung recruitment maneuvers

INTERVENTIONS:
Other: Specific lung recruitment maneuvers — Specific lung recruitment maneuvers will be performed to measure the potential for lung recruitment at different levels of positive end-expiratory pressure (PEEP) provided by the mechanical ventilator. Electrical impedance tomography signals, synchronized signals of airway pressure and flow, esophageal pressure (if available), and volumetric capnography (if available) will be recorded continuously, during the time span of the protocol for offline analysis.

SUMMARY:
The RECRUIT study is a multinational, multicenter physiological observational study conducted by the PLUG working group. It is a single-day study (1.5-2 hours) associated with specific lung (de)recruitment maneuvers to verify the feasibility of measuring the potential for lung recruitment in mechanically ventilated patients with ARDS by electrical impedance tomography (EIT).

DETAILED DESCRIPTION:
Despite higher positive end-expiratory pressure (PEEP) being associated with multiple physiologic benefits, randomized clinical trials comparing higher vs. lower PEEP levels failed to show improved survival of ARDS patients. Higher PEEP should fully exploit its benefits only when implemented in patients with higher potential for alveolar recruitment (i.e., the decrease of non-aerated lung tissue at higher airway pressure) or in patients with airway closure. Retrospective analysis of randomised clinical trials with PEEP suggests that when high PEEP is used in responders (oxygenation), survival may be better. Conversely, in the absence of significant recruitment, higher PEEP should be avoided and lower PEEP might be recommended.

Titration of PEEP provided by the mechanical ventilator in patients with severe lung injury should thus be based on bedside information on lung recruitability. However, no valid method exists to define the best PEEP to optimize recruitment and minimize lung overdistention. Recruitability varies and is often not assessed. Electrical impedance tomography (EIT) is a non-invasive bedside imaging technique for measuring the potential for lung recruitment in ARDS patients. By performing lung (de)recruitment maneuvers and in-depth analyses, we will define lung recruitability indices and develop methods for real-time and personalized PEEP selection. This study will prove the feasibility of minimizing risks associated with inadequate mechanical ventilation by EIT.

ELIGIBILITY:
Inclusion Criteria:

* Intubated moderate and severe ARDS according to the Berlin definition (PaO2/FiO2 ratio <= 200 mmHg)
* Under continuous sedation with or without paralysis

Exclusion Criteria:

* Age <18 years
* Bronchopleural fistula
* Pure COPD exacerbation
* Contraindication to EIT monitoring (e.g. burns, pacemaker, thoracic wounds limiting electrode belt placement)
* Hemodynamic instability (Systolic BP < 75 mmHg or MAP < 60 mmHg despite vasopressors and/or heart rate < 55 bpm)
* Attending physician deems the transient application of high airway pressures to be unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated mechanically ventilated patients will be considered for enrolment in the first week of ARDS diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Potential for lung recruitment | 2 hours
  The potential for lung recruitment will be assessed with EIT. Several methods will be used and compared, based on e.g. pixel information of lung aeration, and pressure-volume characteristics at different PEEP steps.

SECONDARY OUTCOMES:
Recruitment-to-inflation (R/I) ratio | 2 hours
EIT-based optimum PEEP level | 2 hours
PEEP level resulting in end-expiratory transpulmonary pressure between 0 and 2 cmH2O | 2 hours
  For those patients with esophageal pressure measurements available
Organ dysfunction as per the sequential organ failure assessment (SOFA) score | Day 1, 3, 7
  SOFA score min-max: 0-24; a higher score is associated with poor prognosis.
Vital status at ICU discharge, 28 days, and hospital discharge | Through study completion, up to 1 year
  Vital status (death/alive) will be assessed via chart review
Ventilator free days | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (4):
- Faculdade de Medicina da University São Paulo, São Paulo, Brazil
- St. Michael's Hospital, Toronto, Ontario, Canada
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Derived] Jonkman AH, Alcala GC, Pavlovsky B, Roca O, Spadaro S, Scaramuzzo G, Chen L, Dianti J, Sousa MLA, Sklar MC, Piraino T, Ge H, Chen GQ, Zhou JX, Li J, Goligher EC, Costa E, Mancebo J, Mauri T, Amato M, Brochard LJ; Pleural Pressure Working Group (PLUG). Lung Recruitment Assessed by Electrical Impedance Tomography (RECRUIT): A Multicenter Study of COVID-19 Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2023 Jul 1;208(1):25-38. doi: 10.1164/rccm.202212-2300OC. PMID 37097986
- [Derived] Otahal M, Mlcek M, Borges JB, Alcala GC, Hladik D, Kuriscak E, Tejkl L, Amato M, Kittnar O. Prone positioning may increase lung overdistension in COVID-19-induced ARDS. Sci Rep. 2022 Oct 3;12(1):16528. doi: 10.1038/s41598-022-20881-6. PMID 36192569
- [Derived] Mlcek M, Otahal M, Borges JB, Alcala GC, Hladik D, Kuriscak E, Tejkl L, Amato M, Kittnar O. Targeted lateral positioning decreases lung collapse and overdistension in COVID-19-associated ARDS. BMC Pulm Med. 2021 Apr 24;21(1):133. doi: 10.1186/s12890-021-01501-x. PMID 33894747
- See also: Website of the PLUG working group — https://www.plugwgroup.org